CLINICAL TRIAL: NCT04967625
Title: Anti-PD-1 Antibody Sintilimab Combined With Anti-angeogensis Inhibitor Anlotinib in Treatment of Extensive-stage Disease Small Cell Lung Cancer After Failure of First Line Standard Therapy : a Single-arm Prospective Phase II Clinical Study
Brief Title: A Phase II Study of Sintilimab Combined With Anlotinib in Treatment of ED-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-SCLC-01
Record Dates: First submitted 2021-07-15; First posted 2021-07-19 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-03

CONDITIONS: Small Cell Lung Cancer Extensive Stage
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: Anti-PD-1 antibody sintilimab combined With anti-angeogensis inhibitor anlotinib for extensive stage disease small cell lung cancer after failure of first line standard therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab + Anlotinib (Experimental): sintilimab 200mg, IV, d1, Q3W and anlotinib 12mg, PO, QD，d1-14, Q3W; treatment until disease progression, unacceptable toxicity, or death
  Interventions: Drug: Sintilimab; Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Sintilimab — A humanized anti-PD-1 monoclonal antibody
Drug: Anlotinib hydrochloride — A tyrosine kinase inhibitor selectively targeting VEGFR-2

SUMMARY:
This is a the researchers launched, single-center, prospective, open-label, single arm ,Phase II clinical study of Sintilimab combined with anlotinib in patients with extensive-stage disease small-cell lung cancer to evaluate the efficacy and safety.

23 patients are expected to be enrolled in this study.

DETAILED DESCRIPTION:
Subjects will receive sintilimab 200mg, IV, Q3W and anlotinib 12mg, PO, QD，d1-14, Q3W treatment until disease progression, unacceptable toxicity, or death.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18, regardless of gender .
* Histologically or cytologically confirmed small cell lung cancer .
* The time after the end of first-line treatment was less than 6 months .
* Subjects must have measurable diseases as defined in RECIST v1.1 .
* Eastern Cooperative Oncology Group (ECOG) performance status scores are 0-2 .
* Adequate hematologic and end organ function .
* Capable of understanding the trial nature and voluntarily signing the written informed consent form .

Exclusion Criteria:

* Radiographic findings showed that the tumor involved large blood vessels or was poorly demarcated from them .
* Radiographic findings showed significant pulmonary cavitation or necrotizing tumor .
* Active brain metastasis or meningeal metastasis .
* With other malignant tumors in the past 5 years, except cancers that have been cured significantly or can be focally cured, e.g. basosquamous carcinoma of skin, or carcinoma cervix in situ .
* With Interstitial lung disease, including drug- induced Interstitial lung disease or radiation pneumonitis .
* With clinically significant cardiovascular disorder .
* Prior exposure to any immune checkpoint inhibitors, including but not limited to other anti-CTLA-4, anti-PD-1 or anti-PD-L1 antibodies .
* Prior exposure to anti-VEGFR therapy .
* Known hypersensitivity to study drug or any of its excipients .
* Treatment with any other investigational agent or participation in another clinical trial within 4 weeks prior to first administration .
* Other conditions that the investigator thinks unsuitable in this study .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-07-26 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 month
  Objective response rate according to RECIST v1.1

SECONDARY OUTCOMES:
DCR | 12 months
  Disease control rate according to RECIST v1.1
DoR | 12 months
  Duration of response according to RECIST v1.1
PFS | 12 months
  Progression-free survival according to RECIST v1.1
OS | on average of 2 years
  Overall survival
Adverse Event | 12 months
  Evaluation of adverse event rate according to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Guangyuan Lou, Principal Investigator — Zhejiang Cancer Hospital